CLINICAL TRIAL: NCT05406674
Title: Body Surface Area-based vs Concentration-based Dosing of Cisplatin for Hyperthermic Intraperitoneal Chemotherapy (HIPEC) in Women With Advanced Ovarian Cancer
Acronym: CisCon
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N21CCI
Record Dates: First submitted 2022-05-31; First posted 2022-06-06 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: FIGO Stage III Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms | interventions — Cisplatin

STUDY DESIGN:
Intervention Model Description: Patients in Arm A are treated with interval cytoreductive surgery (with no more than 1 cm residual disease) and cispaltin-based HIPEC with a dosage of 100 mg/m2.
  Patients in Arm B are treated with interval cytoreductive surgery (with no more than 1 cm residual disease) and cisplatin- based HIPEC with a dosage of 40 mg/L perfusate.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Active Comparator): Patients in Arm A are treated with interval cytoreductive surgery (with no more than 1 cm residual disease) and cispaltin-based HIPEC with a dosage of 100 mg/m2
  Interventions: Drug: Cisplatin 100 mg/m2
- Arm B (Experimental): Patients in Arm B are treated with interval cytoreductive surgery (with no more than 1 cm residual disease) and cisplatin- based HIPEC with a dosage of 40 mg/L perfusate.
  Interventions: Drug: Cisplatin 40 mg/l

INTERVENTIONS:
Drug: Cisplatin 100 mg/m2 — Cisplatin 100 mg/m2 milligram(s)/square meter
  Other Names: LO1XA; NDC 16729-288; SUB07483MIG; PL 20075/0123
  Arms: Arm A
Drug: Cisplatin 40 mg/l — Cisplatin 40 mg/I milligram(s)/litre
  Other Names: LO1XA; NDC 16729-288; SUB07483MIG; PL 20075/0123
  Arms: Arm B

SUMMARY:
Cytoreductive surgery (CRS) with the addition of hyperthermic intraperitoneal chemotherapy (HIPEC) is used in current clinical practice in selected patients with advanced ovarian cancer. Clinical evidence for the benefit of HIPEC in ovarian cancer comes from the pivotal phase 3 OVHIPEC trial. Worldwide, two established strategies exist for dosing of HIPEC protocols, which follow either a body surface area (BSA)-based or a concentration-based approach. Since both strategies result in different exposure to intra-peritoneal chemotherapy, we aim to compare the pharmacokinetics and safety of both strategies.

ELIGIBILITY:
Inclusion Criteria:

1. signed and written informed consent
2. age ≥ 18 years
3. patients eligible for interval cytoreductive surgery

   1. histological proven FIGO stage III primary high grade serous ovarian, fallopian tube, or extra-ovarian cancer
   2. when only cytology is performed to confirm the diagnosis ovarian carcinoma, immunohistochemistry should be performed including keratin 7, keratin 20, p53, PAX8
   3. neo-adjuvant chemotherapy consists of (at least) 3 courses of carboplatin/paclitaxel
   4. following 2 cycles of chemotherapy no progression should occur
4. treated with optimal or complete interval cytoreductive surgery
5. fit for major surgery, WHO performance status 0-2
6. adequate bone marrow function (hemoglobin level >5.5 mmol/L; leukocytes >3 x 109/L; platelets >100 x 109 /L)
7. adequate hepatic function (ALT, AST and bilirubin <2.5 times upper limit of normal)
8. adequate renal function (creatinine clearance ≥ 60 ml/min using Cockcroft-Gault formula or 24-hour measurement or ml/min/1,73 m2 using MDRD or CKD-EPI)
9. able to understand the patient information

Exclusion Criteria:

1. history of previous malignancy treated with chemotherapy
2. opting for fertility-sparing surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Intratumoral platinum (Pt) concentration at the end of perfusion after 90 minutes (in ng/mg wet tissue) | End of perfusion after 90 minutes

SECONDARY OUTCOMES:
Toxicity evaluation (CTCAE 5.0) | The occurrence of adverse events will be monitored until 6 weeks after surgery
  Grade 3-5 will be reported
Platinum (Pt) concentration in normal tissue (in ng/mg wet tissue) | End of perfusion
Platinum (Pt) concentration in tumor tissue after 30 minutes and 60 minutes of perfusion (in ng/mg wet tissue) | After 30 minutes and 60 minutes of perfusion
Concentration versus time curve and area-under-the-curve (AUC) of intra-peritoneal Platinum (Pt) during perfusion | During perfusion
Maximum Concentration (Cmax) Platinum (Pt) in perfusate during perfusion | During perfusion
Time to Maximum Concentration (Tmax) Platinum (Pt) in perfusate during perfusion | During perfusion
Terminal elimination half-life (t1/2) Platinum (Pt) in perfusate during perfusion | During perfusion
Clearance from perfusate at the end of perfusion | End of perfusion
Overall Survival (OS) | Will be evaluated after 3 and 5 years after the last patient last visit

CONTACTS AND LOCATIONS:
Overall Officials: W. van Driel, MD PhD, Principal Investigator — NKI-AvL
Locations (2):
- Netherlands (2):
  - Antoni van Leeuwenhoek (NKI-AVL), Amsterdam
  - UMCU, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided